CLINICAL TRIAL: NCT01291719
Title: Insulin Balanced Infusion System Control of Glucose
Brief Title: Insulin Balanced Infusion System
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Admetsys Corporation (Industry)
Responsible Party: Principal Investigator, Timothy Valk MD, Chief Scientist, Admetsys Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBIS-1
Record Dates: First submitted 2011-02-05; First posted 2011-02-08 (Estimated); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Hyperglycemia; Diabetes
Keywords: closed loop glucose control; intensive care glucose control
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Insulin and glucose infusion in closed loop control; intervention is glucose control with insulin and glucose infusion
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- insulin and glucose infusion (Experimental): trial of experimental technique in outpatient setting; the group under study will be comprised of type 1 and type 2 diabetic individuals ; they will have automated treatment using algorithm which regulates balancing infusions of glucose and/or insulin intravenously without manual intervention; blood glucose target of 80-180 mg/dl will be guide for the automated system
  Interventions: Device: glucose and insulin infusions

INTERVENTIONS:
Device: glucose and insulin infusions — combined algorithm directed glucose and insulin infusion with 5 minute blood glucose measurements to direct glucose control; regular insulin and glucose are infused intravenously as adjusted by the algorithm without manual intervention in the group of diabetic individuals under study to adjust the glucose level to a target range of 80-180 mg/dl

SUMMARY:
The purpose of this study is to study the use of a counterbalancing system of glucose and insulin infusion with frequent blood glucose monitoring and combined adaptive algorithm can produce tight glycemic control without hypoglycemia; study to develop a closed loop for use in intensive care units and surgery

DETAILED DESCRIPTION:
The study is using an experimental design outpatient with individuals having treatment using an automated closed loop glucose control unit; glucoses are measured every 5 minutes using a intravenous glucose sensor and infusion of glucose and insulin are altered without manual intervention as directed by algorithm

ELIGIBILITY:
Inclusion Criteria:

* type 1 or type 2 diabetic individuals on insulin ages 21-85 with A1c 7-9.9%
* glucose at time of study > 150 mg/dl

Exclusion Criteria:

* pregnancy
* renal or hepatic disease
* corticosteroids
* poor intravenous access
* anemia
* electrolyte abnormality

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-11; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
glucose control in target range | data will be evaluated within 6 months after completion of all 40 studies
  blood glucose measurements in target range (80-125 mg/dl)

SECONDARY OUTCOMES:
hypoglycemia | data will be evaluated within 6 months after all 40 studies are completed
  blood glucose <70 mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Timothy W Valk, MD, Principal Investigator — Admetsys Corporation
Locations (1):
- 3113 Lawton Road, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
with publication the data will be shared

REFERENCES:
- [Result] Hashemi N, Valk T, Houlind K, Ejskjaer N. Insulin-Based Infusion System: Preliminary Study. J Diabetes Sci Technol. 2019 Sep;13(5):935-940. doi: 10.1177/1932296818821349. Epub 2019 Jan 24. PMID 30678470
- [Result] Hashemi N, Valk T, Houlind K, Ejskjaer N. Insulin-Based Infusion System: Advancing the Development. J Diabetes Sci Technol. 2019 Sep;13(5):941-948. doi: 10.1177/1932296819832876. Epub 2019 Mar 10. PMID 30854885